CLINICAL TRIAL: NCT01544634
Title: Evaluation of Any Steroid Sparing Effect of Beta Blocker Therapy on Airway Hyper-responsiveness in Stable, Mild to Moderate Asthmatics
Brief Title: Beta Blocker Therapy in Mild to Moderate Asthmatics
Acronym: ANDA1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Principal Investigator, William J Anderson, Clinical Research Fellow, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011RC16; 2011-002512-89 (EudraCT Number)
Record Dates: First submitted 2012-02-24; First posted 2012-03-06 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Asthma
Keywords: Asthma; Propranolol; Inhaled corticosteroids; Steroid sparing agent; Airway hyper-responsiveness
MeSH Terms: conditions — Asthma; Respiratory Hypersensitivity | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propranolol + Low dose Qvar (Experimental)
  Interventions: Drug: Propranolol; Drug: Qvar 50
- Placebo + high dose Qvar (Active Comparator)
  Interventions: Drug: Placebo; Drug: Qvar 100

INTERVENTIONS:
Drug: Propranolol — Propranolol: 10mg bd for 1 week, 20mg bd for 2 weeks, 80mg MR for 4 weeks.
  Arms: Propranolol + Low dose Qvar
Drug: Placebo — Placebo tablets: 1 tab bd for 2 weeks, 1 tab od for 4 weeks
  Arms: Placebo + high dose Qvar
Drug: Qvar 50 — Qvar 50, 1 puff bd for 6 weeks
  Arms: Propranolol + Low dose Qvar
Drug: Qvar 100 — Qvar 100, 2 puffs bd for 6 weeks
  Arms: Placebo + high dose Qvar

SUMMARY:
Current asthma medicines include inhalers. A common type of inhaler is called a 'beta-agonist' (e.g. salbutamol). They improve asthma symptoms by stimulating areas in the airway causing it to widen. Although these drugs are useful short term, long term use can make asthma worse in some people.

'Beta-blockers' are the complete opposite type of medication. Just now they are avoided in patients with asthma. Beta-blockers cause problems in asthmatics in the short term, including severe asthma attacks.

The other mainstay of inhaler treatment for asthma is inhaled steroid or 'preventer' medication. These work by dampening down the inflammation in the lungs that occurs in asthma.

New research has suggested that longer term use of beta-blockers can also reduce airway inflammation which may improve asthma control. This research was done in asthmatic patients who didn't need inhaled steroids to control their asthma. At the moment the investigators are studying to see if there is a benefit of beta-blocker use for asthma over and above asthmatics own usual doses of inhaled steroids.

In this study, the investigators will be trying to find out if adding a beta blocker to a smaller dose of steroid inhaler has the same effect on asthma control as just using a higher dose of steroid inhaler by itself.

ELIGIBILITY:
Inclusion Criteria:

* Stable mild to moderate asthma
* Histamine PC20 </= 8mg/ml
* Receiving inhaled corticosteroid 0-1000ug daily (BDP equivalent dose)
* FEV1 > 60% predicted
* Diurnal variability < 30%
* Reliever use </= 8puffs/day
* ECG demonstrating sinus rhythm

Exclusion Criteria:

* Uncontrolled symptoms of asthma
* Systolic BP<110mmHg
* Heart rate<60bpm
* Pregnancy or lactation
* Heart block
* Heart rate limiting medications currently prescribed
* Asthma exacerbation within 6 months of study commencement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-04-04 (Actual); Primary Completion 2013-05-25 (Actual); Study Completion 2013-05-25 (Actual)

PRIMARY OUTCOMES:
Change in Histamine provocative concentration causing 20% fall in FEV1 (PC20)at 6 weeks | Change from baseline to 6 weeks
  Measurement of airway hyper-reactivity (a hallmark of asthma).

SECONDARY OUTCOMES:
Change in Impulse oscillometry parameters at 6 weeks | Change from baseline to 6 weeks
  Change in: Resistance at 5Hz, Resistance at 20Hz, Reactance at 5Hz, Frequency of resonance, Area under reactance curve.
Change in Spirometry parameters at 6 weeks | Change from baseline to 6 weeks
  Change in: Forced expiratory volume in 1 second (FEV1); forced vital capacity (FVC); forced expriatory flow between 25-75% of vital capacity; FEV1/FVC ratio.
Change in resting heart rate at 6 weeks | Change from baseline to 6 weeks
  Abosolute change in heart rate at 6 weeks will be a secondary outcome. Participants will measure their own heart rate at home on a daily basis and compare this to a given cut-off value, below which they will be advised to contact a trial doctor.
Change in resting blood pressure at 6 weeks | Change from baseline to 6 weeks
  Blood pressure will be monitored at each visit, or if patients develop symptoms that may be due to low blood pressure.
Change in exhaled tidal nitric oxide levels at 6 weeks | Change from baseline to 6 weeks
Change in overnight urinary cortisol/creatinine ratio (OUCC) at 6 weeks | Change from baseline to 6 weeks
  Systemic effects from inhaled corticosteroids can be measured using OUCC.
Change in symptom scores (Asthma control questionnaire and Asthma quality of life questionnaire) at 6 weeks | Change from baseline to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William J Anderson, MBChB, Principal Investigator — University of Dundee; Brian J Lipworth, MD, Study Director — University of Dundee
Locations (1):
- Asthma and Allergy Research Group, University of Dundee, Dundee, Scotland, United Kingdom

REFERENCES:
- [Background] Morales DR, Guthrie B, Lipworth BJ, Donnan PT, Jackson C. Prescribing of beta-adrenoceptor antagonists in asthma: an observational study. Thorax. 2011 Jun;66(6):502-7. doi: 10.1136/thoraxjnl-2011-200067. Epub 2011 Apr 1. PMID 21459857
- [Background] Lin R, Peng H, Nguyen LP, Dudekula NB, Shardonofsky F, Knoll BJ, Parra S, Bond RA. Changes in beta 2-adrenoceptor and other signaling proteins produced by chronic administration of 'beta-blockers' in a murine asthma model. Pulm Pharmacol Ther. 2008;21(1):115-24. doi: 10.1016/j.pupt.2007.06.003. Epub 2007 Jul 4. PMID 17689122
- [Background] Nguyen LP, Omoluabi O, Parra S, Frieske JM, Clement C, Ammar-Aouchiche Z, Ho SB, Ehre C, Kesimer M, Knoll BJ, Tuvim MJ, Dickey BF, Bond RA. Chronic exposure to beta-blockers attenuates inflammation and mucin content in a murine asthma model. Am J Respir Cell Mol Biol. 2008 Mar;38(3):256-62. doi: 10.1165/rcmb.2007-0279RC. Epub 2007 Dec 20. PMID 18096872
- [Background] Hanania NA, Singh S, El-Wali R, Flashner M, Franklin AE, Garner WJ, Dickey BF, Parra S, Ruoss S, Shardonofsky F, O'Connor BJ, Page C, Bond RA. The safety and effects of the beta-blocker, nadolol, in mild asthma: an open-label pilot study. Pulm Pharmacol Ther. 2008;21(1):134-41. doi: 10.1016/j.pupt.2007.07.002. Epub 2007 Jul 17. PMID 17703976
- [Background] Lipworth BJ, Williamson PA. Think the impossible: beta-blockers for treating asthma. Clin Sci (Lond). 2009 Oct 12;118(2):115-20. doi: 10.1042/CS20090398. PMID 19807697
- [Derived] Anderson WJ, Short PM, Jabbal S, Lipworth BJ. Inhaled corticosteroid dose response in asthma: Should we measure inflammation? Ann Allergy Asthma Immunol. 2017 Feb;118(2):179-185. doi: 10.1016/j.anai.2016.11.018. Epub 2017 Jan 3. PMID 28065396
- [Derived] Anderson WJ, Short PM, Williamson PA, Manoharan A, Lipworth BJ. The inverse agonist propranolol confers no corticosteroid-sparing activity in mild-to-moderate persistent asthma. Clin Sci (Lond). 2014 Dec;127(11):635-43. doi: 10.1042/CS20140249. PMID 24938324